CLINICAL TRIAL: NCT01744106
Title: A Multicenter, Randomized, Placebo-Controlled Study of Pseudoephedrine for the Temporary Relief of Nasal Congestion in Children With the Common Cold
Brief Title: A Multicenter Study of Pseudoephedrine for the Temporary Relief of Nasal Congestion in Children With the Common Cold
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Perrigo Company (Industry)
Collaborators: McNeil Consumer Healthcare Division of McNEIL-PPC, Inc. (Industry); Pfizer (Industry); GlaxoSmithKline (Industry); Chattem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRGO-PSE-09001
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Nasal Congestion Associated With the Common Cold
MeSH Terms: interventions — Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- pseudoephedrine hydrochloride 30 mg tablets (Experimental): Test product
  Interventions: Drug: pseudoephedrine hydrochloride 30 mg tablets
- placebo tablets (Placebo Comparator): Placebo
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: pseudoephedrine hydrochloride 30 mg tablets
  Arms: pseudoephedrine hydrochloride 30 mg tablets
Drug: Placebo tablets
  Arms: placebo tablets

SUMMARY:
This study is designed to confirm the effectiveness of single-ingredient pseudoephedrine in children for the temporary relief of nasal congestion due to the common cold, an indication described under 21 CFR 341.80(b)(1).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, ages 6 through 11 years, are experiencing the common cold, but are otherwise healthy.
2. Subjects have an onset of cold symptoms within the past 2.5 days before screening and are experiencing self-reported nasal congestion of at least stuffy severity (score = 3 or 4).
3. Subjects have at least two of the following additional symptoms due to common cold: runny nose, sneezing, sore throat, headache, body achiness, and cough, as deemed by the parent.
4. Subjects can swallow oral tablets without chewing them (based on a pretest of successfully swallowing a placebo tablet at screening)
5. Findings from the medical history review and vital signs are within the range of clinical acceptability, as determined by the investigator.
6. Subject and legally authorized representative are likely to be compliant and complete the study.
7. Subject's legally authorized representative has signed and dated the informed consent form. Subject has given verbal assent, and has signed and dated the informed assent form.
8. Female subjects who have reached menarche must have a negative urine pregnancy test at screening. These subjects must have practiced abstinence for at least three months prior to study entry and for the duration of the study. A second pregnancy test will be given when the subject returns to the clinic after the last dose.
9. Subject and legally authorized representative can read and understand English.
10. Subject's legally authorized representative who signs informed consent is available to administer all assessments and study medication on days 1 and 2.

Exclusion Criteria:

1. Have any of the following medical conditions: heart disease, high blood pressure, thyroid disease, diabetes, peripheral vascular disease, increased intraocular pressure, prostatic hypertrophy
2. Are under treatment for a hyperexcitability disorder with a medication regimen that has not been stable for at least 3 months
3. Are currently experiencing an asthmatic episode
4. Are experiencing symptoms of seasonal or perennial allergic rhinitis
5. Are currently or within the last 24 hours having symptoms of vomiting or diarrhea
6. Have been exposed to immediate family members with the flu within the past week
7. Are exhibiting signs or symptoms of, or diagnosed with sinusitis, pneumonia, strep throat, acute otitis media, or influenza
8. Are experiencing a fever 103˚F or higher at screening
9. Are from homes where there is smoking in the home around the child.
10. Are currently taking a monoamine oxidase inhibitor (MAOI), or have taken a MAOI within two weeks of screening (e.g., isocarboxazid - Marplan, phenelzine - Nardil, selegiline - Eldepryl, Emsam, Zelapar, and tranylcypromine - Parnate). Note: subjects may not discontinue taking a MAOI solely of the purposes of qualifying for the study.
11. Have a known sensitivity or allergy to pseudoephedrine, phenylephrine, or acetaminophen or any of the excipients of the drug product
12. Have taken any oral cold or allergy medicine within 12 hours of enrollment, or intranasal decongestants within 24 hours of enrollment except for single-ingredient OTC analgesics
13. Have the need to take additional medications, including cough and cold (i.e., oral or intranasal antihistamines, intranasal steroids, intranasal decongestants), or herbal/dietary supplements during the study, with the exception of acetaminophen, a medication regimen for a hyperexcitability disorder that has been stable for at least three months or a daily vitamin or multivitamin/multimineral supplement
14. Have participated in another clinical study within 30 days before entry
15. Have another child from the household currently participating in this study
16. Have a history of drug, alcohol, or tobacco use (older children)
17. Are involved directly or indirectly with the conduct and administration of this study (i.e., children of principal investigator, subinvestigator, study coordinators, other study personnel, employees of Perrigo, and the families of each).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 565 (Actual)
Dates: Start 2012-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Nasal Congestion Severity (NCSi) (instantaneous) scores | 1 Day
  Weighted sum of change from baseline in Nasal Congestion Severity (NCSi) (instantaneous) scores over the first eight hours of treatment on Day 1

SECONDARY OUTCOMES:
change from baseline in NCSi scores from 0 to 4 hours | Day 1
  Sum of change from baseline in NCSi scores from 0 to 4 hours after the first dose on Day 1
change from baseline in NCSi scores from 6, 7, and 8 hours | Day 1
  Weighted sum of change from baseline in NCSi scores from 6, 7, and 8 hours after the first dose on Day 1
Nasal Congestion Relief (NCR) reflective scores at 4 hours and 8 hours | Day 1
  Sum of Nasal Congestion Relief (NCR) reflective scores at 4 hours and 8 hours on Day 1
NCSi score at each time point from 0 to 8 hours | Day 1
  NCSi score at each time point from 0 to 8 hours after the first dose on Day 1
NCSr (reflective) scores at 6 hours and 12 hours | Day 2
  Sum of NCSr (reflective) scores at 6 hours and 12 hours on Day 2
NCSr scores at 6 and 12 hours | Day 2
  NCSr scores at 6 and 12 hours on Day 2

OTHER OUTCOMES:
change from baseline in the Nasal Symptom and Function (NSF) composite score of NCSi | Day 1
  Weighted sum of change from baseline in the Nasal Symptom and Function (NSF) composite score of NCSi, nasal breathing, and nasal clearing over the first eight hours of treatment on Day 1
Sum of change from baseline in NSF composite score from 0 to 4 hours | Day 1
  Sum of change from baseline in NSF composite score from 0 to 4 hours after the first dose on Day 1
Weighted sum of change from baseline in NSF composite score from 6, 7, and 8 hours | Day 1
  Weighted sum of change from baseline in NSF composite score from 6, 7, and 8 hours after the first dose on Day 1
morning sleep score on Days 2 through 7 | Day 7
  Change from baseline in morning sleep score on Days 2 through 7
NSF composite score on Days 2 through 7 | Day 7
  Change from baseline in NSF composite score on Days 2 through 7
NSF + S (sleep) composite score on Days 2 through 7 | Day 7
  Change from baseline in the NSF + S (sleep) composite score on Days 2 through 7

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Emmaus Research Center, Anaheim, California
  - WCCT Global, LLC, Costa Mesa, California
  - Advanced Clinical Research - Boise, Boise, Idaho
  - Bluegrass Clinical Research, Louisville, Kentucky
  - Meridian Clinical Research, Omaha, Nebraska
  - Rapid Medical Research, Cleveland, Ohio
  - Carolina Ear, Nose and Throat Clinic, Orangeburg, South Carolina
  - Meridian Clinical Research - Dakota Dunes, Dakota Dunes, South Dakota
  - ClinPoint Trials, LLC, Waxahachie, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Advanced Clinical Research - West Jordan, West Jordan, Utah